CLINICAL TRIAL: NCT06407479
Title: Comparison of Eccentric Muscle Training and Proprioceptive Neuromuscular Facilitation Techniques in Individuals With Non-specific Neck Pain
Brief Title: Comparison of Eccentric Muscle Training and Proprioceptive Neuromuscular Facilitation Techniques in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar4
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- proprioceptive (Experimental): proprioceptive neuromuscular facilitation technique application
  Interventions: Other: proprioceptive neuromuscular facilitation technique group
- eccentric (Experimental): eccentric muscle training technique application
  Interventions: Other: eccentric muscle training technique application group
- Control (Active Comparator): no intervention group
  Interventions: Other: Control

INTERVENTIONS:
Other: proprioceptive neuromuscular facilitation technique group — Proprioceptive Neuromuscular Facilitation Technique group; In addition to the exercises applied to the participants and the control group, combined isotonic contractions and dynamic stabilization will be used as facilitation techniques, and hold-relax technique will be used as an inhibition technique.
  Arms: proprioceptive
Other: eccentric muscle training technique application group — Eccentric Muscle Training Technique: Participants will receive eccentric muscle training in addition to the exercises given to the control group. Before the application, 5-minute warm-up exercises will be given to the neck area. Eccentric muscle training will be applied to the muscles of the participants in the cervical region. Eccentric exercise will be strengthened in the cervical region muscles in the direction of movement in each plane, that is, flexion / extension and lateral flexion. The movements will first be explained and demonstrated to the patient.
  Arms: eccentric
Other: Control — No intervention will be made.
  Arms: Control

SUMMARY:
It was aimed to compare the eccentric exercise training given to the neck muscles of people with non-specific neck pain and the proprioceptive neuromuscular facilitation (PNF) technique on pain, endurance and functionality.

DETAILED DESCRIPTION:
The study was planned as a quantitative study. Volunteer individuals with nonspecific neck pain between the ages of 18-65 will be included in the study, and the participants will be randomly distributed into 3 groups. Control group (n=15), proprioceptive neuromuscular facilitation technique application group (n=15), eccentric muscle training technique application group (n=15). People included in the study will be explained in detail and will be asked to sign a voluntary consent form approved by the ethics committee. Demographic information of individuals in all three groups will be recorded first. Participants in all three groups will be evaluated at the beginning and end of the applications. In our study, participants were evaluated with the McGill Pain Questionnaire to evaluate the character and character of pain, their physical fitness with the Deep Neck Flexor Endurance Test (DBFET), their functionality related to daily living activities with the Neck Disability Index (NEI), and their quality of life with the World Health Organization Short Form of Quality of Life (WHOYKA-CF). ) Tampa Kinesiophobia Scale (TKÖ) and a goniometer for Cervical Region Joint Range of Motion Measurement will be used to evaluate kinesiophobia, which is the fear of pain and re-injury, as well as anxiety towards activity and physical movement. This study will be planned five times a week for six weeks. Stretching and stabilization exercises will be applied to the control group in 3 sets of 10 repetitions.

ELIGIBILITY:
INCLUSION CRITERIA

* Being between the ages of 18-65
* History of neck pain that has persisted for at least 7 days
* Agreeing to participate in the study
* Having the ability to read and write Turkish. EXCLUSION CRITERIA
* Radiculopathy and structural disorder in the cervical region,
* Surgery to the cervical region,
* Inflammatory disease,
* Severe psychological illness,
* Presence of infection in the bone and soft tissue in the cervical spine,
* Malignancy,
* Advanced osteoporosis,
* Those with upper extremity pathologies,
* Having a neurological disease that will prevent treatment
* Having previously undergone cervical region and spine surgery
* Having been included in a physiotherapy program for the neck and back area in the last 6 months,
* It was defined as the administration of drugs such as NSAIDs (Nonsteroidal Anti-Inflammatory Drugs) and opioids in the last 24 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Cervical Deep Flexor Muscle Endurance Test | 8 weeks
  Patients were asked to lie in a supine position with knees flexed at 90° and hands on the abdomen in a hook position. A 0.5 kilogram (kg) weight was placed on the forehead with the help of a band passed over the ears. The patients were asked to first perform cervical retraction and then 10° cervical flexion, and the degree of flexion was determined with the help of a goniometer. The patients were asked to maintain this position and the time was determined with a stopwatch and recorded in seconds. Patients must be able to maintain this position for 60 seconds (sec) in order to have sufficient muscle endurance. Those below this period have insufficient muscle endurance. Cervical flexion for 60 seconds. Patients holding it above were considered to have sufficient endurance and were not included in the study.
World Health Organization Quality of Life Survey Short Form | 8 weeks
  The scale measures 28 general health, physical, psychological, social and environmental well-being and consists of 26 questions. Turkey version consists of 27 questions. The 27th question is the national question that determines the Environmental Score. Since each domain expresses the quality of life in its own field independently of each other, domain scores are calculated between 4-20. As the score increases, the quality of life increases.
Neck Disability Index | 8 weeks
  Neck Disability Index will be used to evaluate the disability specific to neck pain. The Neck Disability Index has been modified from the Oswestry Disability Index. It consists of 10 sections: pain intensity, personal care, weight bearing, reading, headache, concentration, working, driving, sleep and recreational activities. Each section consists of 6 answers and is scored from 0, no disability, to 5, representing total disability. According to total score; 0-4: no limitation, 5-14: mild limitation, 15-24: moderate limitation, 25-34: severe limitation, 34 and above: completely limited.
Tampa Kinesiophobia Scale | 8 weeks
  Tampa Kinesiophobia Scale was used to evaluate kinesiophobia, which is a state of anxiety that develops against activity and physical movement due to fear of pain and re-injury. It was developed to differentiate between non-excessive fear and phobia in patients with chronic musculoskeletal pain. It is frequently used in the literature to evaluate movement-related fear and anxiety. The scale is a 17-item scale that includes parameters of injury, re-injury and fear-avoidance in work-related activities. As the score increases, it is accepted that the kinesiophobia of the individual with pain increases.Results consist of a total raw score (range between 17 and 68) A low score indicates low kinesiophobia.
Cervical joint goniometric measurements | 8 weeks
  Goniometric measurements in the neck are methods used to evaluate and record neck joint range of motion. These measurements are important to evaluate the patient's condition during the treatment process, follow the progress and create the treatment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra SÖKMEN YILDIRIM, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmgren T, Bjornsson Hallgren H, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. BMJ. 2012 Feb 20;344:e787. doi: 10.1136/bmj.e787. PMID 22349588
- [Background] Heredia-Rizo AM, Petersen KK, Madeleine P, Arendt-Nielsen L. Clinical Outcomes and Central Pain Mechanisms are Improved After Upper Trapezius Eccentric Training in Female Computer Users With Chronic Neck/Shoulder Pain. Clin J Pain. 2019 Jan;35(1):65-76. doi: 10.1097/AJP.0000000000000656. PMID 30222615
- [Background] Espi-Lopez GV, Aguilar-Rodriguez M, Zarzoso M, Serra-Ano P, Martinez DE LA Fuente JM, Ingles M, Marques-Sule E. Efficacy of a proprioceptive exercise program in patients with nonspecific neck pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2021 Jun;57(3):397-405. doi: 10.23736/S1973-9087.20.06302-9. Epub 2020 Oct 13. PMID 33047944
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Gillani SN, Ain Q-, Rehman SU, Masood T. Effects of eccentric muscle energy technique versus static stretching exercises in the management of cervical dysfunction in upper cross syndrome: a randomized control trial. J Pak Med Assoc. 2020 Mar;70(3):394-398. doi: 10.5455/JPMA.300417. PMID 32207413